CLINICAL TRIAL: NCT02308007
Title: Solubilized Metronidazole And/oR Terconazole Gels Intra-Vaginal Efficacy and Safety
Brief Title: Multi-Center Study of New Medications to Treat Vaginal Infections
Acronym: SMART GIVES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Curatek Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTC-001 (Trial 3)
Record Dates: First submitted 2014-12-01; First posted 2014-12-04 (Estimated); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Vaginal Infection
MeSH Terms: conditions — Vaginitis | interventions — terconazole; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Terconazole vaginal gel (Active Comparator): One applicator full at bedtime
  Interventions: Drug: Terconazole
- Metronidazole vaginal gel (Active Comparator): One applicator full at bedtime
  Interventions: Drug: Metronidazole
- Terconazole/metronidazole vaginal gel (Active Comparator): One applicator full at bedtime
  Interventions: Drug: Terconazole/metronidazole

INTERVENTIONS:
Drug: Terconazole
  Arms: Terconazole vaginal gel
Drug: Metronidazole
  Arms: Metronidazole vaginal gel
Drug: Terconazole/metronidazole
  Arms: Terconazole/metronidazole vaginal gel

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of terconazole/metronidazole gel in the treatment of vaginal infections

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of vaginal infection that is confirmed by laboratory testing and:
* Capable of providing written informed consent or assent
* Currently not menstruating and not anticipating menses during treatment
* If heterosexually active, subject must be post-menopausal for ≥ 1 year, surgically sterile, or practicing an acceptable form of birth control
* Negative pregnancy test
* Other criteria as identified in the protocol

Exclusion Criteria:

* Other infectious causes of vulvovaginitis
* Subject has recently used, or is expected to require the concomitant use of prohibited medications/products
* Nursing mother
* Use of any investigational drug within 30 days of enrollment
* History of hypersensitivity to any ingredient/component of the formulations
* Other criteria as identified in the protocol

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Borgman, Ph.D., Study Director — Curatek Pharmaceuticals
Locations (51):
- United States (51):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama
  - Precision Trials, AZ, Phoenix, Arizona
  - MomDoc Womens Health Research, Scottsdale, Arizona
  - DelSol Research, Tucson, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Gossmont Center for Clinical Research, La Mesa, California
  - Genesis Center for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Downtown Women's Health Care, Denver, Colorado
  - Red Rocks Ob/Gyn, Lakewood, Colorado
  - Women's Health CT Ob/Gyn, Bridgeport, Connecticut
  - Precision Clinical Research, Coral Springs, Florida
  - KO Clinical Research, LLC, Fort Lauderdale, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Discovery Clinical Research, Plantation, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Georgia Regents University, Augusta, Georgia
  - Atlanta North Gynecology, Roswell, Georgia
  - Mount Vernon CLinical Research, Sandy Springs, Georgia
  - Rosemark Womens Care Specialists, Idaho Falls, Idaho
  - Women's Health Practice, Champaign, Illinois
  - Indiana University, Indianapolis, Indiana
  - Praetorian Pharmaceutical Research, LLC, Marrero, Louisiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Women Under Study, New Orleans, Louisiana
  - Wayne State University, Detroit, Michigan
  - Women's Healthcare Specialists, PC, Kalamazoo, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Clinic of Lincoln, Lincoln, Nebraska
  - Legacy Women's Health, Las Vegas, Nevada
  - R. Garn Mabey Jr., MD Gynecology, Las Vegas, Nevada
  - Lawrence Ob/Gyn Clinical Research LLC, Lawrenceville, New Jersey
  - Women's Health Research Center, Plainsboro, New Jersey
  - Suffolk OB/GYN, Port Jefferson, New York
  - East Carolina Women's Center, New Bern, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Radiant Research, Columbus, Ohio
  - Complete Healthcare for Women, Columbus, Ohio
  - Drexel University, Philadelphia, Pennsylvania
  - Philapelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Magnolia Ob/Gyn Research Center, Myrtle Beach, South Carolina
  - James T. Martin, MD, North Charleston, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Discovery Clinical Trials, Dallas, Texas
  - Signature Gyn Services, Fort Worth, Texas
  - Texas Children's Hospital for Women, Houston, Texas
  - TMC Life Research, Inc., Houston, Texas
  - Harborview Medical Center, Seattle, Washington
  - Women's Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Terconazole Vaginal Gel: One applicator full at bedtime
  Terconazole
- Metronidazole Vaginal Gel: One applicator full at bedtime
  Metronidazole
- Terconazole/Metronidazole Vaginal Gel: One applicator full at bedtime
  Terconazole/metronidazole
Period: Overall Study
Arm/Group | Terconazole Vaginal Gel | Metronidazole Vaginal Gel | Terconazole/Metronidazole Vaginal Gel
Started | 159 | 159 | 157
Completed | 83 | 84 | 82
Not Completed | 76 | 75 | 75
Not completed — Normal Gram stain or neg yeast culture | 66 | 64 | 67
Not completed — Positive for STD at Baseline | 7 | 11 | 7
Not completed — Lost to Follow-up | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: modified intent-to-treat (mITT) population includes all subjects randomized to treatment and administered at least one dose of study drug. In addition, subjects must have a Nugent score of 4 or more on Baseline visit Gram stain slide and a Baseline visit yeast culture positive for Candida species.
Groups:
- Total: Total of all reporting groups
Arm/Group | Terconazole Vaginal Gel | Metronidazole Vaginal Gel | Terconazole/Metronidazole Vaginal Gel | Total
Number analyzed (Participants) | 83 | 84 | 82 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (9.17) | 31.0 (9.43) | 32.6 (10.57) | 31.7 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 84 | 82 | 249
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 9 | 39
  Not Hispanic or Latino | 68 | 69 | 73 | 210
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 52 | 54 | 50 | 156
  White | 30 | 26 | 28 | 84
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 83 | 84 | 82 | 249

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure of Mixed Infection (BV and VVC) as Assessed by the Investigator at the Test-of-cure Visit
Description: The percentage of participants with clinical cure of both bacterial vaginosis (BV) AND vulvovaginal candidiasis (VVC) was compared between the combination therapy and the two single entity treatments. Clinical cure of BV is defined as: discharge has returned to normal/physiologic, negative whiff test, and saline wet mount is <20% clue cells. Clinical cure of VVC is defined as resolution of all signs and symptoms attributable to vulvovaginal candidiasis
Time Frame: 7-14 days after beginning treatment
Population: mITT population (Baseline Nugent Gram stain score of 4 or more, and positive baseline yeast culture, and used at least one dose of study medication)
Measure: Count of Participants; unit: Participants
Arm/Group | Terconazole Vaginal Gel | Metronidazole Vaginal Gel | Terconazole/Metronidazole Vaginal Gel
Number analyzed (Participants) | 83 | 84 | 82
Participants | 31 | 29 | 43
Statistical Analysis 1: Comparison: Metronidazole Vaginal Gel vs Terconazole/Metronidazole Vaginal Gel; Test type: Superiority; p = 0.030, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Terconazole Vaginal Gel vs Terconazole/Metronidazole Vaginal Gel; Test type: Superiority; p = 0.073, Chi-squared, Corrected
Statistical Analysis 3: Comparison: Metronidazole Vaginal Gel vs Terconazole/Metronidazole Vaginal Gel; Stratified by race (black, white, or other race); Test type: Superiority; p = 0.0204, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Terconazole Vaginal Gel vs Terconazole/Metronidazole Vaginal Gel; Stratified by race (black, white, or other race); Test type: Superiority; p = 0.0493, Cochran-Mantel-Haenszel

2. Secondary Outcome: Cure of the BV Component of Mixed Infection
Description: The percentage of participants with both BV and VVC who had clinical cure of bacterial vaginosis (BV) was compared between the combination therapy and the two single entity treatments. Clinical cure of BV was defined as: 1. discharge has returned to normal/physiologic, 2. the whiff test is negative for any amine "fishy" odor, 3. the saline wet mount is <20% clue cells
Time Frame: 7-14 days after beginning treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Terconazole Vaginal Gel | Metronidazole Vaginal Gel | Terconazole/Metronidazole Vaginal Gel
Number analyzed (Participants) | 83 | 84 | 82
Participants | 38 | 46 | 54
Statistical Analysis 1: Comparison: Terconazole Vaginal Gel vs Terconazole/Metronidazole Vaginal Gel; Test type: Superiority; p = 0.015, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Metronidazole Vaginal Gel vs Terconazole/Metronidazole Vaginal Gel; Difference for Terconazole/metronidazole vaginal gel cures minus metronidazole vaginal gel cures; Test type: Superiority; p = 0.193, Chi-squared, Corrected

3. Secondary Outcome: Cure of the VVC Component of Mixed Infection
Description: The percentage of participants with both BV and VVC who had clinical cure of VVC was compared between the combination therapy and the two single entity treatments.Clinical cure of VVC was defined as complete resolution of all signs and symptoms attributable to VVC
Time Frame: 7-14 days after beginning treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Terconazole Vaginal Gel | Metronidazole Vaginal Gel | Terconazole/Metronidazole Vaginal Gel
Number analyzed (Participants) | 83 | 84 | 82
Participants | 52 | 37 | 53
Statistical Analysis 1: Comparison: Metronidazole Vaginal Gel vs Terconazole/Metronidazole Vaginal Gel; Test type: Superiority; p = 0.012, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Terconazole Vaginal Gel vs Terconazole/Metronidazole Vaginal Gel; Test type: Superiority; p = 0.918, Chi-squared, Corrected

4. Secondary Outcome: Microbiologic and Mycologic Cure
Description: The percentage of participants with both microbiologic and mycologic cure was compared between the combination therapy and the two single entity treatments. Yeast cultures were performed and Gram stains of vaginal fluid were graded according to Nugent's criteria. Microbiologic cure requires normal Nugent gram stain score and mycologic cure requires negative yeast culture.
Time Frame: 7-14 days after beginning treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Terconazole Vaginal Gel | Metronidazole Vaginal Gel | Terconazole/Metronidazole Vaginal Gel
Number analyzed (Participants) | 83 | 84 | 82
Participants | 19 | 5 | 24

5. Secondary Outcome: Number of Participants Reporting Complete Resolution of Symptoms by Test of Cure Visit
Description: Subjects reported if symptoms completely resolved and the date of resolution. The percentage of participants reporting complete resolution of symptoms was compared between arms.
Time Frame: 7-14 days after beginning treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Terconazole Vaginal Gel | Metronidazole Vaginal Gel | Terconazole/Metronidazole Vaginal Gel
Number analyzed (Participants) | 83 | 84 | 82
Participants | 49 | 44 | 49

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Adverse events were collected at study visits, from subject diaries and from spontaneous reports
Time Frame: Any time during study participation (up to 30 days)
Population: Safety population, defined as all subjects randomized to treatment and administered at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Terconazole Vaginal Gel | Metronidazole Vaginal Gel | Terconazole/Metronidazole Vaginal Gel
Number analyzed (Participants) | 149 | 151 | 154
Participants | 44 | 40 | 44

ADVERSE EVENTS:
Time Frame: The safety population includes all participants randomized to treatment and administered at least one dose of study drug, and includes subjects who had a negative yeast culture and/or normal gram stain at the baseline visit. Adverse events were collected over the entire course of the study (up to 30 days after beginning treatment).
Description: Adverse events were collected through direct questioning at each post-baseline visit, by participant diaries, and by spontaneous reporting.
Arm/Group | Terconazole Vaginal Gel | Metronidazole Vaginal Gel | Terconazole/Metronidazole Vaginal Gel
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/151 | 0/154
Serious Adverse Events (participants affected / at risk) | 1/149 | 0/151 | 0/154
Other Adverse Events (participants affected / at risk) | 5/149 | 6/151 | 8/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terconazole Vaginal Gel (N=149) | Metronidazole Vaginal Gel (N=151) | Terconazole/Metronidazole Vaginal Gel (N=154)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terconazole Vaginal Gel (N=149) | Metronidazole Vaginal Gel (N=151) | Terconazole/Metronidazole Vaginal Gel (N=154)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 5 (5) | 6 (6) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators have the right to disclose and publish results of the Study conducted by them; provided that, in order to protect any Curatek confidential information, Investigator shall submit to Curatek manuscripts at least 30 days before submission for publication or 10 days before public presentation. After that time, Investigator is free to submit the manuscript for publication or deliver the presentation, provided Investigator removes any confidential information as directed by Curatek.

DOCUMENTS (2):
  • Study Protocol (2015-03-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT02308007/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT02308007/SAP_001.pdf